CLINICAL TRIAL: NCT05854355
Title: Reducing Sedentary Behaviour and Promoting Physical Activity in Children Aged 7-9 Years: Developing, Feasibility and Pilot Testing a Low-cost, Multi-component, School-based Classroom Intervention.
Brief Title: Children- Sit Less, Move More (C-SLAMM): Increasing Physical Activity and Decreasing Sedentary Behaviour in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Northern Ireland Chest Heart and Stroke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REC.21.0027
Record Dates: First submitted 2023-03-30; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Physical Inactivity; Sedentary Behavior; Health Behavior; Child Behavior; Physical Activity
MeSH Terms: conditions — Sedentary Behavior; Health Behavior; Child Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: Four schools allocated to receive the intervention; four schools allocated to the control group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group received the multi-component school and home-based intervention (physical activity programme (aimed to increase children's physical activity and decrease sedentary behaviour)
  Interventions: Other: C-SLAMM Study
- Control (No Intervention): The primary school children in the control group did not receive the intervention.
  The control arm continued with their usual practice and lesson delivery, no environmental changes were made to their classrooms.

INTERVENTIONS:
Other: C-SLAMM Study — The intervention arm includes using innovative behavioural, pedagogical, and environmental strategies within the classroom, school, and home settings to get children moving more and sitting less. The strategies were based on strategies used in Transform-Us! involved incorporating movement into everyday class lessons - the delivery of the lesson changes, not the content. Resources included health lessons, active lessons, active breaks, active homework to do with parents, active environments, and newsletters for parents.
  Arms: Intervention

SUMMARY:
The Children Sit Less, Move More (C-SLAMM) study aims to test the feasibility and potential effect of a multi-component school and home-based pilot cluster randomized control trial on reducing sedentary behavior and increasing physical activity in children.

This pilot intervention will be an 8-week two-armed cluster RCT. Individuals (children aged 7-9 years) will be the unit of analysis and schools (cluster) randomly assigned to one of two arms: (1) Physical activity and sedentary behavior (intervention arm), or (2) current practice (control arm). The design conduct and reporting of the intervention with adhere to the Consolidation Standards of Reporting Trials (CONSORT) guidelines and is guided by the Standard Protocol Items for Randomized Trials (SPIRIT) Statement.

DETAILED DESCRIPTION:
The C-SLAMM study is an 8-week school-and home-based feasibility, two-armed pilot cluster randomized controlled trial.

A convenience sample of primary schools in Northern Ireland will be invited to take part in the study. Baseline measurements will proceed randomization, and an identical set of measures will be taken from participants in week 8 of the intervention.

Individuals (Primary 4 and Primary 5 children, aged 7-9 years) will be the unit of analysis and schools (clusters) will be randomly assigned to one of two conditions: (1) intervention condition or (2) current practice (control condition). Given the nature of the intervention, blinding of schools and participants will not be possible following randomization. The researcher responsible for subsequent data collection and analysis will not be blinded to group allocation. Any differences between the intervention and control groups will be by chance and adjusted for in the analyses. Schools randomized to control will be offered information on the intervention and associated materials at the end of the intervention.

The intervention is, adapted from the previously tested Transform-Us! trial and informed by a qualitative study was on the perceived barriers and facilitators of physical activity within the classroom, school and/or home environment (REC/20/0033).

The C-SLAMM study will use innovative behavioral, pedological, and environmental strategies within the classroom, school, and home settings to get children moving more and sitting less. Resources include health lessons, active lessons, active breaks, active homework to do with parents, active environments, and newsletters for parents. Each week teachers will be advised to incorporate elements of the intervention within the classroom setting. Teachers will modify the delivery of at least one class lesson per week (~30 minutes) so that children will complete the lesson standing up. Teachers will be provided with a suite of standing lesson delivery methods that can be modified to any class topic. In addition, every two-hour classroom teaching block will be interrupted every 30 minutes with a 2-minute guided light-intensity activity break. This will equate to a total of six minutes interrupted sitting time every two hours. Furthermore, each class will be provided with six standing desks so that children can rotate learning activities at 'standing stations'. A novelty timer will be given to each class so that teachers can monitor 2-minute standing breaks and every 30-minutes of sitting class time.

To compare the effects of the intervention against usual practice, schools assigned to the control arm will be requested to continue with their usual practice and lesson delivery, no environmental changes will be made to their classrooms. The participants in the control schools will be asked to complete the same study measurements as those in the intervention schools at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Primary school pupil
* Year 4 (Key Stage 1) or Year 5 (Key Stage 2)
* 7-9 years
* Living in Northern Ireland

Exclusion Criteria:

* Cannot speak English
* Severe psychological or neurological condition

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 162 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
Sitting time (mins) | 7 days at baseline and at follow-up (8 weeks)
  Change in time spent sitting using activPAL inclinometer device

SECONDARY OUTCOMES:
Standing time (mins) | 7 days at baseline and at follow-up (8 weeks)
  Change in time spent standing using activPAL inclinometer device
Stepping time (mins) | 7 days at baseline and at follow-up (8 weeks)
  Change in time spent stepping using activPAL inclinometer device
Steps | 7 days at baseline and at follow-up (8 weeks)
  Changes in Steps using activPAL inclinometer device
Sit to stand transitions | 7 days at baseline and at follow-up (8 weeks)
  Changes in Sit to stand transitions using activPAL inclinometer device
Height (m) | 7 days at baseline and at follow-up (8 weeks)
  Change in height measured with portable Stadiometer
Weight (kg) | 7 days at baseline and at follow-up (8 weeks)
  Change in weight measured with electronic weighing scales
Body Mass index (kg/m2) | 7 days at baseline and at follow-up (8 weeks)
  Change in BMI calculated from height and weight measures

CONTACTS AND LOCATIONS:
Overall Officials: Marie Murphy, PhD, Principal Investigator — University of Ulster
Locations (1):
- Ulster University, Newtownabbey, Co. Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nally S, Carlin A, Gallagher AM, Wilson JJ, Lahart IM, Salmon J, Murphy MH. The Children - Sit Less, Move More (C-SLAMM) pilot intervention: Feasibility and acceptability of a multi-component school and home-based intervention to promote physical activity. PLoS One. 2025 Nov 19;20(11):e0335933. doi: 10.1371/journal.pone.0335933. eCollection 2025. PMID 41259385